CLINICAL TRIAL: NCT03715816
Title: Work Breaks During Minimally Invasive Surgery - Target-group Specific Development of Work Break Schedules
Brief Title: Work Breaks During Simulated Minimally Invasive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Tessy Luger, Principal Investigator, University Hospital Tuebingen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UKT-2018AS0-1835
Record Dates: First submitted 2018-09-26; First posted 2018-10-23 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Work-break Schedules
Keywords: endoscopy; minimally invasive surgery; passive breaks; active breaks; muscle activity; back curvature

STUDY DESIGN:
Masking Description: The study is not blinded, because the subject(s) will know which of the three experimental conditions they are exposed to (control without breaks; intervention with passive or active breaks). The same applies to the experimenter(s).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No breaks (No Intervention): Subjects will simulate a 90-min laparoscopic activities in the laboratory.
- Passive breaks (Experimental): Subjects will simulate a 90-min laparoscopic activities in the laboratory, and after 30 and 60 min of work, they will be provided a 2.5-min break during which they can have a rest.
  Interventions: Behavioral: Work break schedule
- Active breaks (Experimental): Subjects will simulate a 90-min laparoscopic activities in the laboratory, and after 30 and 60 min of work, they will be provided a 2.5-min break during which they will be performing some mobilisation exercises for the back, shoulder, and neck.
  Interventions: Behavioral: Work break schedule

INTERVENTIONS:
Behavioral: Work break schedule — Participants will receive 2.5-min breaks during a 90-min simulated laparoscopic surgery in the laboratory. The breaks will be either passive (simple rest) or active (selected mobilization exercises).
  Other Names: passive break; active break
  Arms: Active breaks; Passive breaks

SUMMARY:
Minimally invasive surgeons have a prevalence of work-related musculoskeletal complaints of up to 86% due to the exposure to static loading, awkward postures, work pressure, and patient's wellbeing. Researchers have developed postural interventions to counteract the prevalence of musculoskeletal complaints and disorders, such as robot-assisted surgeries, arm-support systems, and rotatable handle pieces. An alternative intervention is to implement work breaks during the surgeries, which has shown to give promising results including that surgery duration does not prolong.

The aim of the current study is to simulate 90-min laparoscopic surgery activities in the laboratory and compare two intervention situations with the control situation. The control situation is without work breaks. The two intervention situations include 2.5-min breaks provided two times, i.e. after every 30-min work period, which are passive (rest) or active (targeted mobilization exercises). The assessment is based on changes in muscular activity on the back and upper extremities, back and upper extremity postures, feelings of discomfort, and work performance.

ELIGIBILITY:
Inclusion Criteria:

* (Student) surgeons, who are familiar with laparoscopic procedures and / or simulated laparoscopic procedures;
* Be able to perform the Peg-Transfer task (Simulab, Seattle, WA, USA) within 3 minutes;
* The participant will give her/his voluntary informed consent after receiving oral and written information of the content and goal of the study.

Exclusion Criteria:

* (Student) surgeons who are not familiar with laparoscopic procedures and / or simulated laparoscopic procedures;
* Not able to perform the Peg-Transfer task within 3 minutes;
* People under the influence of intoxicants, analgesics, or muscle relaxants;
* Alcohol abuse;
* People with cardiovascular diseases;
* People with a heart pacemaker;
* People with a disability who, due to their restriction at a workplace of this kind, will not be able to participate;
* People with Diabetes Mellitus;
* People with severe muscle contractions of the lower extremities, back or arms;
* People with acute ailments or pain, which make(s) them unable to participate;
* People who are unable to complete the examination program due to language or cognitive obstacles;
* Depending on the degree of severity, people with diseases of the veins and joints of the lower extremities, spine, muscle disorders, symptomatic neurological-psychiatric diseases, acute pain syndromes, maladies or other current diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Rating of perceived discomfort | Change from baseline (0 min) to directly after (90 min) each experimental condition
  Discomfort will be assessed using an 11-point numeric rating scale, ranging from 0 (no discomfort at all) to 10 (maximally imaginable discomfort). It will be assessed directly before and directly after each experimental condition.

SECONDARY OUTCOMES:
Root-mean-square of electrical muscle activity recordings using electromyography | Average root-mean-square of muscle activity over the time period running from baseline (0 min) to directly after (90 min) each experimental condition
  Selected target muscles in the arms (deltoid acromialis, extensor digitorum, flexor carpi radialis), shoulder (trapezius descendens) and back (erector spinae lumbalis) will be continuously recorded with electromyography. From the electromyographic signal, the root-mean-square will be calculated and averaged over the time period in each experimental condition.
Median power frequency of electrical muscle activity recordings using electromyography | Average median power frequency f muscle activity over the time period running from baseline (0 min) to directly after (90 min) each experimental condition
  Selected target muscles in the arms (deltoid acromialis, extensor digitorum, flexor carpi radialis), shoulder (trapezius descendens) and back (erector spinae lumbalis) will be continuously recorded with electromyography. From the electromyographic signal, the median power frequency will be calculated and averaged over the time period in each experimental condition.
Posture of the spine / back | Average posture over time period baseline (0 min) to end (90 min) of each experimental condition
  Using gravimetric position sensors, the curvature of the back will be recorded as well as the head position and movement with respect to the trunk. Recordings are continuous and average angles (kyphosis, lordosis, neck angle) will be calculated per time period.
Heart rate | Average heart activity over time period baseline (0 min) to end (90 min) of each experimental condition
  Continuous recording electrocardiography allows calculating the heart rate, a parameter reflecting the central stress state of the participant. The average heart rate will be calculated per time period.
Work performance | Change from baseline (0 min) to directly after (90 min) each experimental condition
  Using the Peg-Transfer Board (Simulab, Seattle, WA, USA), subjects will perform this task for exaclty 1 minute. Time is recorded after one repetition is finished and final performance for the overall minute is recorded as well.
Workload | Assessed at 90 min, directly after each experimental condition
  Using the Hart and Staveland's NASA Task Load Index (TLX) method, workload is assessed for 6 dimensions where participants put a cross on one of the 21 lines on the 21-point scales, which range from left (very satisfied; way too much; much to short; clearly increased) to right (very unsatisfied; way too few; much to long; clearly reduced).
Participant evaluation | Assessed at 90 min, directly after the experimental conditions with intervention
  Self-developed questionnaire assessing aspects of applicability and acceptability of the tested interventions in the field. All questions will be multiple choice questions, resulting in categorical variables (scales ranging from 1 [very satisfied / true] to 4 [very unsatisfied / not true]).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Occupational and Social Medicine and Health Services Research, University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luger T, Rieger MA, Bonsch R, Kramer B, Seibt R, Steinhilber B. Active and passive work breaks during simulated laparoscopy among laparoscopic surgeons: study protocol for a controlled, randomised cross-over laboratory trial. BMJ Open. 2020 Nov 19;10(11):e038952. doi: 10.1136/bmjopen-2020-038952. PMID 33444192
- [Derived] Luger T, Bonsch R, Seibt R, Kramer B, Rieger MA, Steinhilber B. Intraoperative active and passive breaks during minimally invasive surgery influence upper extremity physical strain and physical stress response-A controlled, randomized cross-over, laboratory trial. Surg Endosc. 2023 Aug;37(8):5975-5988. doi: 10.1007/s00464-023-10042-9. Epub 2023 Apr 21. PMID 37084097
- See also: Homepage of the responsible Institute — https://www.medizin.uni-tuebingen.de/de/das-klinikum/einrichtungen/institute/arbeitsmedizin-sozialmedizin-und-versorgungsforschung
- See also: Page 285: poster presentation with preliminary results presented at the PREMUS 2019 conference in Bologna, Italy — http://www.premus2019.com/wp-content/uploads/2019/09/PREMUS-2019-Abstact-30.08.19.pdf